CLINICAL TRIAL: NCT04640909
Title: Impact of Treatment With Targeted Therapies on the Generation of Effective CAR T Cells in Patients With Chronic Lymphocytic Leukemia
Brief Title: Impact of Treatment With Targeted Therapies on the Generation of CAR T Cells in CLL Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CLL2020
Record Dates: First submitted 2020-11-09; First posted 2020-11-23 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-10

CONDITIONS: CLL; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR T Cells generation (Other): CAR T Cells generation at baseline and after 6 and 12 months of treatment
  Interventions: Other: Peripheral blood samples withdrawal

INTERVENTIONS:
Other: Peripheral blood samples withdrawal — Peripheral blood samples evaluation

SUMMARY:
In this biological study, blood samples will be collected from patients with CLL treated with targeted agents (ibrutinib and venetoclax) to assess the impact of these treatments on the generation of CAR T cells in terms of manufacturing efficiency, immunophenotypic characteristics and functional properties.

DETAILED DESCRIPTION:
This is a biological study aimed at analyzing the features of CAR T cells generated in CLL patients treated with ibrutinib or venetoclax.

To this purpose, blood samples will be collected from patients with CLL before starting therapy with ibrutinib or venetoclax and after 6 and 12 months of treatment.

Anti-CD19 CAR T cells will be generated and tested for: (i) viability, expansion and generation efficiency; (ii) phenotypic characteristics, in terms of CD4/CD8 composition, differentiation subset distribution, exhaustion markers and expression of immune checkpoint molecules; (iii) in vitro functional properties, in terms of proliferation ability, cytokines production, cytotoxic activity and killing of target cells. CAR T cells produced from the same patient at different timepoints will be compared. Phenotypic and functional data on CAR T cells will be also correlated with main CLL prognostic factors (e.g. IGHV mutational status, FISH abnormalities, TP53 mutation status) and outcome variables (response status, duration of response).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLL/SLL meeting the IWCLL 2008 criteria;
* ≥18 years old;
* Indication for treatment with targeted therapies (i.e. ibrutinib or venetoclax);
* Anticipated possibility to collect blood samples at the baseline and at 6- and 12-month timepoints;
* Signed written informed consent according to ICH/EU/GCP and national local laws;
* Confirmed availability of the laboratory to enroll and to process patient samples.

Exclusion Criteria:

* Expected treatment duration with targeted drug < 12 months, according to treating physician;
* Previously treated with more than 2 lines of CLL-directed therapy;
* Concurrent use of systemic steroids or chronic use of immunosuppressive medications;
* Active HBV (HBsAg+ or HBV DNA+) or HCV or HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Cell killing rate of anti-CD19 CAR T cells | After 12 months of treatment
  Assessment of the cytotoxic functions of anti-CD19 CAR T cells generated from CLL patients in terms of cell killing rate before and during treatment with targeted agents (i.e. ibrutinib or venetoclax).

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Irccs Ospedale S. Raffaele - Milano - Unità Neoplasie Linfocitarie B, Milan
  - Aou Città Della Salute E Della Scienza, Ospedale S. Giovanni Battista Molinette - Torino - Sc Ematologia - Università Degli Studi Di Torino, Torino